CLINICAL TRIAL: NCT01099865
Title: High-sensitivity C-reactive Protein and UKPDS Risk Score in Type 2 Diabetes: Nalysis With 18F-Fluorodeoxyglucose Positron Emission Tomography
Brief Title: High-sensitivity C-reactive Protein and United Kingdom Prospective Diabetes Study (UKPDS) Risk Score in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Korea Unoiversity Guro Hospital, IRB
Other Study IDs: PET(DM)
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Atherosclerosis; Type 2 Diabetes
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The UKPDS risk score is recommended to assess global risk for future coronary heart disease (CHD) events in primary prevention. Recently, high-sensitivity C-reactive protein (hsCRP) has emerged as a strong independent risk factor for CHD. 18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) is a promising imaging technique for the evaluation of vascular inflammation that reflects vulnerable atherosclerotic plaque.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes

Exclusion Criteria:

* Myocardial infarction, unstable angina, stroke, peripheral artery disease, or cardiovascular revascularization
* Resting blood pressure ≥160/100 mmHg
* Malignancy, or severe renal or hepatic disease
* Participants were free of any lipid-lowering therapies and postmenopausal hormone replacement therapy at least the 6 month period prior to enrollment
* History of inflammatory condition or those taking medications that might affect inflammatory status within 6 months

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital Dept. of Endocrinology, Seoul, South Korea